CLINICAL TRIAL: NCT05556031
Title: The Reduction of Decompensation and Unnecessary Cardiac Failure Emergency Admissions: Ambulatory Heart Failure Service Model
Brief Title: Ambulatory Heart Failure Service Model Study
Acronym: REDUCE-HF
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Other Study IDs: 2022.245
Record Dates: First submitted 2022-09-15; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- REDUCE: Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — Standard clinical care

SUMMARY:
The aim of the study is to assess the efficacy of this new ambulatory service model in reducing heart failure hospitalization (HHF), improving clinical as well as functional outcomes of post-discharge patients with Heart Failure of reduced ejection fraction (HFrEF) and Heart failure with preserved Ejection Fraction (HFpEF).

ELIGIBILITY:
Inclusion Criteria:

* Dyspnoea (exertional or at rest) and 2 of the following signs:
* Congestion on chest X-ray
* Rales on chest auscultation
* Clinically relevant oedema (e.g. ≥1+ on a 0 to 3+ scale)
* Elevated jugular venous pressure
* NT-proBNP ≥300 pg/mL (Patients with AF: NT-proBNP ≥900 pg/mL)
* Heart failure hospitalization that requires the treatment of a minimum single dose of 40 mg of i.v. furosemide (or equivalent i.v loop diuretics)
* Ambulatory patients

Exclusion Criteria:

* Cardiogenic shock required inotropics
* Cardiac mechanical support implantation like LVAD
* Life expectancy less than 1 year due to underlying significant comorbidities like metastatic cancer or end-stage COPD
* Haemodynamically severe uncorrected primary cardiac valvular disease planned for surgery or intervention during the course of the study.
* End stage renal failure or eGFR <15 mL/min/1.73m2 as measured during index hospitalization or requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with heart failure with preserved ejection fraction (HFpEF, EF > 50%) and heart failure with reduced ejection fraction (HFrEF, EF <50%)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 90 days
  A composite of all-cause mortality, number of heart failure events (including hospitalization for heart failure (HHF), urgent heart failure visits and unplanned outpatient visits), time to first heart failure event will be aggregated to evaluate overall clinical outcome

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ-TSS) | 1 year
  Change from baseline in KCCQ-TSS, higher score reflects better outcome, Maximum score 100.
NT-proBNP level | 1 year
  Change from baseline in NT-proBNP level
Risk of Heart failure | 1 year
  Change in NYHA class, ELAN-HF score, and MAGGIC Risk score. and Seattle Heart Failure Model Risk Prediction
Change in overall Cardiac function | 90 days
  Evaluated by left ventricular ejection fraction (LVEF), left ventricle volume index, global longitudinal strain (GLS), E/E' ratio, left atrial (LA) volume index and LA GLS, inferior vena cava (IVC) size, right ventricular systolic pressure (RVSP) and functional mitral regurgitation (MR) will be aggregated to represent the overall cardiac function
Major Adverse Cardiovascular Event | 1 year
  Time to first occurrence of cardiovascular death or heart failure event
Hypertensive heart failure (HHF) | 90 days after initial hospital discharge
  Occurrence of HHF
Quality adjusted Life years gained | 1 year
  Cost effectiveness of ambulatory heart failure service for heart failure events avoided and quality adjusted life years (QALY) gained.
Change in 6 minute hall walk (6MHW) | 90 days
  Change in 6 minute hall walk (6MHW) result compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No